CLINICAL TRIAL: NCT03550378
Title: A Phase 2a, Randomised, Double-Blind, Placebo-Controlled Study to Evaluate the Efficacy, Safety, and Pharmacokinetics of MEDI0382 in Subjects With Type 2 Diabetes Mellitus and Renal Impairment
Brief Title: A Study to Look at the Effect MEDI0382 Has on Blood Sugar in People With Type 2 Diabetes and Kidney Problems and Also to Check That MEDI0382 is Well Tolerated
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: MedImmune LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: D5670C00013; 2018-000019-26 (EudraCT Number)
Record Dates: First submitted 2018-04-27; First posted 2018-06-08 (Actual); Results first posted 2020-04-13 (Actual); Last update posted 2020-04-13 (Actual); Status verified 2020-03

CONDITIONS: Type II Diabetes Mellitus; Renal Insufficiency
Keywords: Type 2 Diabetes Mellitus; MEDI0382; Renal Impairment; Glucose concentration; Hemoglobin A1c
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Renal Insufficiency | interventions — cotadutide

STUDY DESIGN:
Intervention Model Description: Randomised, Double-Blind, Placebo-Controlled
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MEDI0382 (Experimental): Participants will receive subcutaneous (SC) dose of MEDI0382 titrated from 50 μg upto 300 μg (50 μg once daily for 4 days, followed by 100 μg daily for 7 days, 200 μg daily for 7 days, and 300 μg daily for 14 days) for 32 days.
  Interventions: Drug: MEDI0382
- Placebo (Placebo Comparator): Participants will receive SC dose of placebo matched to MEDI0382 once daily for 32 days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: MEDI0382 — Participants will receive subcutaneous MEDI0382 titrated from 50 μg upto 300 μg (50 μg once daily for 4 days, followed by 100 μg daily for 7 days, 200 μg daily for 7 days, and 300 μg daily for 14 days) for 32 days.
  Arms: MEDI0382
Drug: Placebo — Participants will receive SC placebo matched to MEDI0382 once daily for 32 days.
  Arms: Placebo

SUMMARY:
A study to look at the effect MEDI0382 has on blood sugar in people with type 2 diabetes and kidney problems and also to check that MEDI0382 is well tolerated.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 and < 85 years at screening.
2. Signed and dated written informed consent (with the exception of consent for genetic and nongenetic research) prior to performing any protocol-related procedures, including screening evaluations.
3. Diagnosed with type 2 diabetes mellitus (T2DM) with glucose control managed with any insulin and/or oral therapy combination where no significant dose changes of oral therapy of more than 50% have occurred in the 3 months prior to screening
4. Body mass index (BMI) between 25 and 45 kg/m^2 (inclusive) at screening
5. Haemoglobin A1c (HbA1c) range of 6.5 % to 10.5% (inclusive) at screening
6. Renal impairment with estimated glomerular filtration rate (eGFR) ≥ 30 and < 60 mL/min/1.73 m^2 at screening. Approximately 16 participants (40%) are required to have a screening eGFR ≥30 and < 45 mL/min/1.73 m^2 and at least 16 participants (40%) are required to have screening eGFR ≥45 and < 60 mL/min/1.73 m^2.
7. Females of childbearing potential must have a negative pregnancy test at screening and randomisation, and must not be lactating. Women of childbearing potential who are sexually active with a non-sterilized male partner must be using at least one highly effective method of contraception from screening and up to 4 weeks after the last dose study drug.

Exclusion Criteria:

1. History or presence of significant medical or psychological conditions, including substance dependence/abuse, or significant abnormalities in laboratory parameters or vital signs including electrocardiogram (ECG), which in the opinion of the investigator, would compromise the participant's safety or successful participation in the study. As an example, severe anaemia (haemoglobin < 7.0 g/dL) could be exclusionary due to blood sampling required by the protocol, at the discretion of investigator.
2. Concurrent participation in another interventional study of any kind and repeat randomisation in this study is prohibited.
3. Any participant who has received another study drug as part of a clinical study or a glucagon-like peptide-1 (GLP-1) analogue-containing preparation within the last 30 days or 5 half-lives of the drug (if known; whichever is longer) at the time of Visit 2.
4. Any participant who has received any of the following medications within the specified timeframe prior to the start of the study (Visit 2)

   * Herbal preparations within 1 week prior to the start of dosing (Visit 4) or drugs licensed for control of body weight or appetite (eg, orlistat, bupropion-naltrexone, phentermine-topiramate, phentermine, lorcaserin) within 30 days (or 5 half-lives of the drug) prior to the start of dosing (Visit 4)
   * Aspirin (acetylsalicylic acid) at a dose greater than 150 mg once daily and within the last 3 days prior to the start of the run-in period (Visit 2)
   * Paracetamol (acetaminophen) or paracetamol-containing preparations at a total daily dose of greater than 3000 mg and within the last 3 days prior to the start of the run-in period (Visit 2)
   * Ascorbic acid (vitamin C) supplements at a total daily dose of greater than 1000 mg and within the last 3 days prior to the start of the run-in period (Visit 2)
   * Opiates, domperidone, metoclopramide, or other drugs known to alter gastric emptying and within 2 weeks prior to the start of dosing (Visit 4)
5. Severe allergy/hypersensitivity to any of the proposed study treatments or excipients
6. Symptoms of acutely decompensated blood glucose control (eg, thirst, polyuria, weight loss), a history of type 1 diabetes mellitus or diabetic ketoacidosis
7. Participants who have undergone a renal transplant
8. Participants with suspicion of acute or subacute renal function deterioration (eg, participants with large fluctuations of creatinine values documented within the 6 months prior to screening)
9. Significant inflammatory bowel disease, gastroparesis, or other severe disease or surgery affecting the upper gastrointestinal (GI) tract including weight-reducing surgery and procedures) which may affect gastric emptying or could affect the interpretation of safety and tolerability data
10. History of acute or chronic pancreatitis
11. Significant hepatic disease (except for non-alcoholic steatohepatitis or nonalcoholic fatty liver disease without portal hypertension or cirrhosis) and/or participants with any of the following results:

    * Aspartate transaminase (AST) ≥ 3 × upper limit of normal (ULN)
    * Alanine transaminase (ALT) ≥ 3 × ULN
    * Total bilirubin ≥ 2 × ULN
12. Poorly controlled hypertension defined as:

    * Systolic blood pressure (BP) > 180 mm Hg
    * Diastolic BP ≥ 100 mm Hg Participants who fail BP screening criteria may be considered for 24-hour ambulatory blood pressure monitoring (ABPM) at the discretion of the investigator. Participants who maintain a mean 24-hour systolic BP ≤ 180 or diastolic BP < 100 mm Hg with a preserved nocturnal dip of > 15% will be considered eligible
13. Unstable angina pectoris, myocardial infarction, transient ischemic attack or stroke within 3 months prior to screening, or participants who have undergone percutaneous coronary intervention or a coronary artery bypass graft within the past 6 months or who are due to undergo these procedures at the time of screening
14. Severe congestive heart failure (New York Heart Association Class III or IV)
15. Basal calcitonin level > 50 ng/L at screening or history/family history of medullary thyroid carcinoma or multiple endocrine neoplasia
16. History of neoplastic disease within 5 years prior to screening, except for adequately treated basal cell skin cancer, squamous cell skin cancer, or in situ cervical cancer
17. Any positive results for serum hepatitis B surface antigen (HBsAg), hepatitis C antibody, and human immunodeficiency virus (HIV) antibody
18. Nephrotic range proteinuria defined as spot urine albumin creatinine ratio (ACR) > 250 mg/mmol at screening
19. History of substance dependence, alcohol abuse, or excessive alcohol intake (defined as an average weekly intake of > 21 alcoholic drinks for men or > 10 alcoholic drinks for women) within 3 years prior to screening, and/or a positive screen for drugs of abuse or alcohol at screening or on Day -5. Participants who use tricyclic antidepressants or benzodiazepines for an established clinical indication may be permitted to enter the study based upon the judgement of the investigator

Ages: 18 Years to 84 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2018-06-29 (Actual); Primary Completion 2019-02-04 (Actual); Study Completion 2019-02-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (6):
- Germany (4):
  - Research Site, Berlin
  - Research Site, Magdeburg
  - Research Site, München
  - Research Site, Münster
- United Kingdom (2):
  - Research Site, Dundee
  - Research Site, Edinburgh

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool. Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- [Derived] Natale P, Green SC, Tunnicliffe DJ, Pellegrino G, Toyama T, Strippoli GF. Glucagon-like peptide 1 (GLP-1) receptor agonists for people with chronic kidney disease and diabetes. Cochrane Database Syst Rev. 2025 Feb 18;2(2):CD015849. doi: 10.1002/14651858.CD015849.pub2. PMID 39963952
- [Derived] Parker VER, Hoang T, Schlichthaar H, Gibb FW, Wenzel B, Posch MG, Rose L, Chang YT, Petrone M, Hansen L, Ambery P, Jermutus L, Heerspink HJL, McCrimmon RJ. Efficacy and safety of cotadutide, a dual glucagon-like peptide-1 and glucagon receptor agonist, in a randomized phase 2a study of patients with type 2 diabetes and chronic kidney disease. Diabetes Obes Metab. 2022 Jul;24(7):1360-1369. doi: 10.1111/dom.14712. Epub 2022 Apr 25. PMID 35403793
- See also: D5670C00013 CSP redacted — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D5670C00013&attachmentIdentifier=1045860c-2e58-48f1-9900-046596519846&fileName=D5670C00013-amendment-4_Redacted.pdf&versionIdentifier=
- See also: D5670C00013 - SAP_Redacted — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D5670C00013&attachmentIdentifier=fbade528-c567-45fe-b186-3c6712adac53&fileName=D5670C00013_-_Statistical_Analysis_Plan_Redacted.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted in the United Kingdom and Germany between 29Jun2018 and 04Feb2019.
Pre-assignment Details: A total of 41 participants were randomized to the study.
Groups:
- Placebo: Participants received subcutaneous dose (SC) of placebo matched to MEDI0382 once daily for 32 days.
- MEDI0382: Participants received SC dose of MEDI0382 titrated from 50 μg upto 300 μg (50 μg once daily for 4 days, followed by 100 μg daily for 7 days, 200 μg daily for 7 days, and 300 μg daily for 14 days) for 32 days.
Period: Overall Study
Arm/Group | Placebo | MEDI0382
Started | 20 | 21
Completed | 20 | 20
Not Completed | 0 | 1
Not completed — Death | 0 | 1

BASELINE CHARACTERISTICS:
Population: As-treated population included all participants who received any dose of study drug and analyzed according to the treatment they actually received.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | MEDI0382 | Total
Number analyzed (Participants) | 20 | 21 | 41
Age, Continuous [Mean (Standard Deviation); unit: Years] | 70.9 (4.7) | 71.1 (7.4) | 71.0 (6.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 9 | 20
  Male | 9 | 12 | 21
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 20 | 21 | 41
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 0 | 0 | 0
  White | 20 | 20 | 40
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline in Plasma Glucose Area Under the Concentration Time-curve From Time 0 to 4 Hours (AUC0-4 Hrs) as Measured by Mixed-meal Tolerance Test (MMTT) to Day 32
Description: The MMTT involved the consumption of a standardised liquid meal (a nutritional supplement containing the components of fat, carbohydrate, and protein, which make up a standard MMTT) within 15 minutes, and timed serial blood samples obtained for measurement of glucose and parameters related to glucose metabolism through 240 minutes after consumption of the standardized meal (with no additional food intake during this time).
Time Frame: Zero minutes before and 15, 30, 45, 60, 90, 120, 180, and 240 minutes after consumption of the standardised meal on Day -5 (Baseline) and Day 32
Population: Intent-to-treat (ITT) population included all participants who received any dose of study drug and analyzed according to their randomized treatment group. Here, "N" signifies only the participants with available data were analyzed for the outcome measure.
Measure: Least Squares Mean (90% Confidence Interval); unit: Percent change in plasma glucose
Arm/Group | Placebo | MEDI0382
Number analyzed (Participants) | 20 | 18
Percent change in plasma glucose | 3.678 [-3.793 to 11.149] | -26.706 [-34.584 to -18.828]
Statistical Analysis 1: Comparison: Placebo vs MEDI0382; Test type: Superiority; p < 0.001, ANCOVA; LS Mean Difference = -30.384, 90% CI 2-sided [-41.270 to -19.498]

2. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs) and Treatment-emergent Serious Adverse Events (TESAEs)
Description: An adverse event (AE) is any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. A serious adverse event (SAE) is an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. The TEAEs are defined as events present at baseline that worsened in intensity after administration of study drug or events absent at baseline that emerged after administration of study drug.
Time Frame: Day 1 through Day 60
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | MEDI0382
Number analyzed (Participants) | 20 | 21
Participants
  TEAEs | 13 | 20
  TESAEs | 2 | 2

3. Secondary Outcome: Number of Participants With Abnormal Vital Signs Reported as TEAEs
Description: Number of participants with abnormal vital signs reported as TEAEs is reported. Vital sign measurements were obtained after the participant had rested in the supine position for at least 10 minutes at the recording time. Abnormal vital signs is defined as any abnormal finding in the vital sign parameters (blood pressure, pulse rate, body temperature, and respiratory rate).
Time Frame: Day 1 through Day 60
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | MEDI0382
Number analyzed (Participants) | 20 | 21
Participants | 0 | 0

4. Secondary Outcome: Change From Baseline in Postural Blood Pressure
Description: The change difference is the change from Day 1 to Day 32 in the difference between systolic blood pressure (SBP) or diastolic blood pressure (DBP) values in standing and supine positions. For this outcome measure, participants with difference (standing-supine) in DBP or SBP on Day 1 and Day 32 were analyzed. For few participants either DBP or SBP was recorded eg, standing DBP was not recorded on Day 1 for 2 participants in Placebo arm and 1 participant in MEDI0382 arm; standing SBP was not recorded on Day 32 for a participant in the Placebo arm.
Time Frame: Baseline (Day 1) through Day 32
Population: As-treated population included all participants who received any dose of study drug and analyzed according to the treatment they actually received. Participants with difference (standing-supine) in DBP or SBP on Day 1 and the participants with difference (standing-supine) in DBP or SBP on Day 32 were analyzed.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Placebo | MEDI0382
Number analyzed (Participants) | 20 | 21
mmHg
  Systolic Blood Pressure: number analyzed (Participants) | 17 | 18
  Systolic Blood Pressure | 0.1 (9.3) | 8.9 (14.2)
  Diastolic Blood Pressure: number analyzed (Participants) | 17 | 17
  Diastolic Blood Pressure | 1.8 (6.3) | 0.8 (5.2)

5. Secondary Outcome: Number of Participants With Abnormal Electrocardiograms (ECGs) Reported as TEAEs
Description: Number of participants with abnormal ECGs reported as TEAEs is reported. Abnormal ECGs is defined as any abnormal findings in heart rate, RR interval, PR interval, QRS, axis, ST-T morphology, and QT intervals from the primary lead of the digital 12-lead ECG.
Time Frame: Day 1 through Day 60
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | MEDI0382
Number analyzed (Participants) | 20 | 21
Participants
  Bradyarrhythmia | 1 | 0
  Bundle branch block left | 1 | 0
  Bundle branch block right | 0 | 1

6. Secondary Outcome: Number of Participants With Abnormal Clinical Laboratory Parameters Reported as TEAEs
Description: Number of participants with abnormal clinical laboratory parameters reported as TEAEs is reported. Abnormal clinical laboratory parameters defined as any abnormal finding during analysis of serum chemistry, hematology, and urine.
Time Frame: Day 1 through Day 60
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | MEDI0382
Number analyzed (Participants) | 20 | 21
Participants
  Hypoglycaemia | 1 | 3
  Alanine aminotransferase increased | 1 | 0
  Aspartate aminotransferase increased | 1 | 0
  Glomerular filtration rate decreased | 0 | 1

7. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events of Special Interest (TEAESIs)
Description: An adverse event of special interest (AESI) was one of scientific and medical interest specific to understanding of the study drug and may require close monitoring and rapid communication by the investigator to the sponsor.
Time Frame: Day 1 through Day 60
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | MEDI0382
Number analyzed (Participants) | 20 | 21
Participants | 0 | 0

8. Secondary Outcome: Change From Baseline in Mean 24-hrs Pulse Rate to the End of Each Dosing Level
Description: Change from baseline in mean 24-hrs pulse rate to the end of each dosing levels: Day 5 for 50 μg; Day 12 for 100 μg, Day 19 for 200 μg, and Day 32 for 300 μg.
Time Frame: Day -5 (Baseline) and on Days 5, 12, 19, and 32
Population: As-treated population included all participants who received any dose of study drug and analyzed according to the treatment they actually received. Here, "n" signifies only the participants with available data were analyzed for the specified time points.
Measure: Mean (Standard Deviation); unit: Beats/min
Arm/Group | Placebo | MEDI0382
Number analyzed (Participants) | 20 | 21
Beats/min
  Day 5: number analyzed (Participants) | 12 | 13
  Day 5 | -0.73 (4.13) | 6.40 (5.53)
  Day 12: number analyzed (Participants) | 11 | 12
  Day 12 | 1.04 (5.07) | 9.01 (7.73)
  Day 19: number analyzed (Participants) | 14 | 13
  Day 19 | 1.32 (5.28) | 12.72 (8.93)
  Day 32: number analyzed (Participants) | 11 | 10
  Day 32 | -0.92 (4.51) | 11.85 (8.82)

9. Secondary Outcome: Change From Baseline in Mean 24-hrs Systolic and Diastolic Blood Pressure to the End of Each Dosing Level
Description: Change from baseline in mean 24-hrs systolic and diastolic blood pressure to the end of each dosing levels: Day 5 for 50 μg, Day 12 for 100 μg, Day 19 for 200 μg, and Day 32 for 300 μg.
Time Frame: Day -5 (Baseline) and on Days 5, 12, 19, and 32
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Placebo | MEDI0382
Number analyzed (Participants) | 20 | 21
mmHg
  Day 5: Systolic Blood Pressure: number analyzed (Participants) | 12 | 13
  Day 5: Systolic Blood Pressure | -3.11 (9.97) | -1.69 (9.06)
  Day 12: Systolic Blood Pressure: number analyzed (Participants) | 11 | 12
  Day 12: Systolic Blood Pressure | -2.67 (12.30) | -4.34 (11.46)
  Day 19: Systolic Blood Pressure: number analyzed (Participants) | 14 | 13
  Day 19: Systolic Blood Pressure | -3.56 (10.15) | -4.72 (11.65)
  Day 32: Systolic Blood Pressure: number analyzed (Participants) | 11 | 10
  Day 32: Systolic Blood Pressure | 2.21 (7.24) | -1.15 (18.43)
  Day 5: Diastolic Blood Pressure: number analyzed (Participants) | 12 | 13
  Day 5: Diastolic Blood Pressure | -0.07 (3.19) | 1.15 (3.64)
  Day 12: Diastolic Blood Pressure: number analyzed (Participants) | 11 | 12
  Day 12: Diastolic Blood Pressure | -0.55 (5.17) | 1.28 (5.22)
  Day 19: Diastolic Blood Pressure: number analyzed (Participants) | 14 | 13
  Day 19: Diastolic Blood Pressure | -0.44 (3.85) | 0.76 (3.75)
  Day 32: Diastolic Blood Pressure: number analyzed (Participants) | 11 | 10
  Day 32: Diastolic Blood Pressure | 1.84 (1.79) | 2.54 (5.34)

10. Secondary Outcome: Change From Baseline in Haemoglobin A1c (HbA1c) to Day 32
Description: Change from baseline in haemoglobin A1c (HbA1c) is reported.
Time Frame: Day 1 (Baseline) and Day 32
Population: as for outcome 1
Measure: Least Squares Mean (90% Confidence Interval); unit: Percent
Arm/Group | Placebo | MEDI0382
Number analyzed (Participants) | 20 | 19
Percent | 0.01 [-0.15 to 0.17] | -0.65 [-0.82 to -0.49]

11. Secondary Outcome: Change From Baseline in Fasting Glucose to Day 32
Description: Change from baseline in fasting glucose is reported.
Time Frame: Day 1 (Baseline) and Day 32
Population: An ITT population included all participants who received any dose of study drug and analyzed according to their randomized treatment group. Here, "N" signifies only the participants with available data were analyzed for the outcome measure.
Measure: Least Squares Mean (90% Confidence Interval); unit: mg/dL
Arm/Group | Placebo | MEDI0382
Number analyzed (Participants) | 20 | 19
mg/dL | 0.60 [-12.89 to 14.08] | -19.55 [-33.39 to -5.71]

12. Secondary Outcome: Change From Baseline in Percentage of Time Spent Within a Target Glucose Range Over a 7-day Period to the Final Week of Treatment
Description: Change from baseline in percentage of time spent within a target glucose range over a 7-day period to the final week of treatment is reported. Target glucose range was considered as 70 mg/dL (3.9 mmol/L) to 180 mg/dL (10 mmol/L).
Time Frame: Baseline (Days -8 to -2), Days 5 to 11, Days 12 to 18, Days 19 to 25, and Days 26 to 32 (final week of treatment)
Population: An ITT population included all participants who received any dose of study drug and analyzed according to their randomized treatment group. Here, "n" signifies only the participants with available data were analyzed for the specified time points.
Measure: Least Squares Mean (90% Confidence Interval); unit: Percentage of time
Arm/Group | Placebo | MEDI0382
Number analyzed (Participants) | 20 | 21
Percentage of time
  Days 5 - 11: number analyzed (Participants) | 17 | 19
  Days 5 - 11 | -10.49 [-20.77 to -0.20] | 12.25 [2.52 to 21.98]
  Days 12 - 18: number analyzed (Participants) | 18 | 19
  Days 12 - 18 | -5.34 [-12.77 to 2.10] | 15.62 [8.39 to 22.86]
  Days 19 - 25: number analyzed (Participants) | 18 | 18
  Days 19 - 25 | -16.05 [-25.02 to -7.08] | 19.18 [10.21 to 28.15]
  Days 26 - 32: number analyzed (Participants) | 18 | 17
  Days 26 - 32 | -21.23 [-33.13 to -9.32] | 14.79 [2.54 to 27.04]

13. Secondary Outcome: Percent Change Frome Baseline in Body Weight to Day 33
Description: Percent change from baseline in body weight is reported.
Time Frame: Day 1 (Baseline) and Day 33
Population: as for outcome 11
Measure: Least Squares Mean (90% Confidence Interval); unit: Percent change in body weight
Arm/Group | Placebo | MEDI0382
Number analyzed (Participants) | 20 | 19
Percent change in body weight | -0.21 [-1.05 to 0.62] | -3.69 [-4.55 to -2.83]

14. Secondary Outcome: Change From Baseline in Absolute Body Weight to Day 33
Description: Change from baseline in absolute body weight is reported.
Time Frame: Day 1 (Baseline) and Day 33
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: Kg
Arm/Group | Placebo | MEDI0382
Number analyzed (Participants) | 20 | 19
Kg | -0.15 (1.84) | -3.39 (2.16)

15. Secondary Outcome: Area Under the Plasma Concentration Time Curve Over a Dosing Duration (AUCτ) of MEDI0382 at 300 μg
Description: Area under the plasma concentration time curve over a dosing duration (AUCτ) of MEDI0382 at 300 μg is reported.
Time Frame: Predose and at 0.5, 1, 2, 4, 6, 8, and 24 hrs postdose on Day 32
Population: Pharmacokinetic (PK) population included all participants who received at least 1 dose of study drug and had at least one PK sample collected with a value above the lower limit of quantitation.
Measure: Geometric Mean (Full Range); unit: ng.hr/mL
Arm/Group | MEDI0382
Number analyzed (Participants) | 16
ng.hr/mL | 285.93 [124.08 to 669.17]

16. Secondary Outcome: Maximum Observed Serum Concentration (Cmax) of MEDI0382 at 300 μg
Description: Maximum observed serum concentration (Cmax) of MEDI0382 at 300 μg is reported.
Time Frame: Predose and at 0.5, 1, 2, 4, 6, 8, and 24 hrs postdose on Day 32
Population: The PK population included all participants who received at least 1 dose of study drug and had at least one PK sample collected with a value above the lower limit of quantitation.
Measure: Geometric Mean (Full Range); unit: ng/mL
Arm/Group | MEDI0382
Number analyzed (Participants) | 18
ng/mL | 16.93 [5.17 to 35.4]

17. Secondary Outcome: Time to Observed Maximum Serum Concentration (Tmax) of MEDI0382 at 300 μg
Description: Time to observed maximum serum concentration (Tmax) of MEDI0382 at 300 μg is reported.
Time Frame: Predose and at 0.5, 1, 2, 4, 6, 8, and 24 hrs postdose on Day 32
Population: as for outcome 16
Measure: Median (Full Range); unit: Hours
Arm/Group | MEDI0382
Number analyzed (Participants) | 18
Hours | 5.6 [4 to 24]

18. Secondary Outcome: Trough Plasma Concentration (Ctrough) of MEDI0382
Description: Trough concentration is the lowest concentration reached by a drug before the next dose is administered. Trough plasma concentration of MEDI0382 is reported.
Time Frame: Days 1, 5, 12, and 19: Predose; and Day 32: Predose and at 0.5, 1, 2, 4, 6, 8, and 24 hrs postdose (Day 33)
Population: The PK population included all participants who received at least 1 dose of study drug and had at least one PK sample collected with a value above the lower limit of quantitation. Here, "n" signifies only the participants with available data were analyzed for the specified time points.
Measure: Geometric Mean (Full Range); unit: ng/mL
Arm/Group | MEDI0382
Number analyzed (Participants) | 21
ng/mL
  Day 1: number analyzed (Participants) | 0
  Day 5: number analyzed (Participants) | 19
  Day 5 | 1.44 [0.48 to 2.58]
  Day 12: number analyzed (Participants) | 19
  Day 12 | 2.03 [0.63 to 3.75]
  Day 19: number analyzed (Participants) | 20
  Day 19 | 3.68 [0.59 to 8.86]
  Day 32: number analyzed (Participants) | 17
  Day 32 | 5.86 [1.3 to 19.4]
  Day 33: number analyzed (Participants) | 19
  Day 33 | 5.96 [2.43 to 19.2]

19. Secondary Outcome: Number of Participants With Positive Anti-drug Antibodies (ADA) Titre to MEDI0382
Description: Number of participants with positive Anti-drug antibodies (ADA) Titre to MEDI0382 is reported.
Time Frame: Pre-dose on Days 1, 12, and 32 and on Day 60
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | MEDI0382
Number analyzed (Participants) | 20 | 21
Participants
  Positive at baseline | 0 | 0
  Positive post-baseline | 0 | 2
  Positive at baseline and post-baseline | 0 | 0
  Not detected at baseline; positive post-baseline | 0 | 2
  Positive at baseline; not detected post-baseline | 0 | 0

ADVERSE EVENTS:
Time Frame: Day 1 through Day 60
Arm/Group | Placebo | MEDI0382
All-Cause Mortality (participants affected / at risk) | 0/20 | 1/21
Serious Adverse Events (participants affected / at risk) | 2/20 | 2/21
Other Adverse Events (participants affected / at risk) | 13/20 | 19/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=20) | MEDI0382 (N=21)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Carotid artery stenosis (Nervous system disorders) | 1 (1) | 0 (0)
Hypertensive crisis (Vascular disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 1 (2) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=20) | MEDI0382 (N=21)
Bradyarrhythmia (Cardiac disorders) | 1 (1) | 0 (0)
Bundle branch block left (Cardiac disorders) | 1 (1) | 0 (0)
Bundle branch block right (Cardiac disorders) | 0 (0) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Vertigo positional (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 5 (5)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 5 (6)
Eructation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Flatulence (Gastrointestinal disorders) | 0 (0) | 2 (2)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 4 (4) | 9 (19)
Vomiting (Gastrointestinal disorders) | 1 (1) | 6 (18)
Complication associated with device (General disorders) | 0 (0) | 1 (1)
Injection site erythema (General disorders) | 0 (0) | 1 (1)
Injection site pruritus (General disorders) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 2 (2) | 3 (3)
Otitis media (Infections and infestations) | 0 (0) | 1 (1)
Pyelonephritis (Infections and infestations) | 1 (1) | 0 (0)
Rhinitis (Infections and infestations) | 2 (2) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Face injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Glomerular filtration rate decreased (Investigations) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 3 (3)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 3 (8)
Hypoglycaemia unawareness (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Carotid artery stenosis (Nervous system disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 2 (2)
Headache (Nervous system disorders) | 2 (3) | 2 (3)
Nervousness (Psychiatric disorders) | 1 (1) | 0 (0)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Night sweats (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin fissures (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin swelling (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
MedImmune has 60 days to review results communications prior to public release and may delete information that compromises on going studies or is considered proprietary. This restriction is not intended to compromise the objective scientific integrity of the manuscript, it being understood that results shall be published regardless of outcome.

DOCUMENTS (2):
  • Study Protocol (2018-11-12): https://cdn.clinicaltrials.gov/large-docs/78/NCT03550378/Prot_000.pdf
  • Statistical Analysis Plan (2018-06-08): https://cdn.clinicaltrials.gov/large-docs/78/NCT03550378/SAP_001.pdf